CLINICAL TRIAL: NCT06791148
Title: Low-dose Radiotherapy Combined With Albumin-bound Paclitaxel and AK112 as Second-line Treatment in Patients With Advanced Gastric or Gastroesophageal Junction（G.GEJ）Cancer Who Failed First-line Therapy：a Single，Phase II Trial
Brief Title: Low-dose Radiotherapy Combined With Chemotherapy and AK112 as Second-line Treatment in Patients With Advanced G/GEJ Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jia Wei, MD, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-C-M-0003
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Radiotherapy; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low-dose radiotherapy plus chemo and AK112 (Experimental): Radiation therapy for metastatic lesions: Radiation therapy begins within 24 hours before medication administration, with a dose of 2Gy per fraction, administered once every three weeks, for a total of four fractions.
  Chemo：albumin-bound paclitaxel ，100-120mg/m2,i.v.,d2,d9,q3w； AK112：20mg/kg, i.v., d2, q3w
  Interventions: Radiation: Low-dose radiotherapy; Drug: albumin-bound paclitaxel; Drug: AK112

INTERVENTIONS:
Radiation: Low-dose radiotherapy — 2Gy/f，q3w，×4f
Drug: albumin-bound paclitaxel — 100-120mg/m2,i.v.,d2,d9,q3w
Drug: AK112 — 20mg/kg, i.v., d2, q3w

SUMMARY:
The study aims to evaluate the efficacy and safety of the combination of albumin-bound paclitaxel and AK112 with low-dose radiotherapy in patients with gastric adenocarcinoma and gastroesophageal junction adenocarcinoma who have failed first-line standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form.
2. ≥18 years and ≤75 years .
3. Histologically confirmed unresectable locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma (AJCC 8.0);failed first-line standard treatment.
4. PS 0-2.
5. Expected survival ≥ 6 months.
6. With at least one measurable lesion (RECIST 1.1 criteria) in the subject .
7. Within 7 days before starting study treatment, no blood components or growth factors have been used, and Adequate organ function is determined by the following criteria:

   Absolute Neutrophil Count (ANC) ≥ 1.5 x 10^9/L;Platelets ≥ 90 x 10^9/L

   ;Hemoglobin ≥ 80 g/L;Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 times ULN; Serum creatinine ≤ 1.5 times ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥ 60 ml/min; Good coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN Cardiac enzyme levels within normal range (minor lab abnormalities deemed not clinically significant by the investigator are allowed)
8. For women of childbearing potential, a negative urine or serum pregnancy test must be obtained within 3 days before the first dose of study drug. If the urine test is inconclusive, a blood pregnancy test is required. Postmenopausal women are defined as those who have had no menses for at least 1 year or have undergone surgical sterilization or hysterectomy.
9. All participants with fertility potential must use contraception with a failure rate <1% during treatment and for 120 days after the last dose of study drug (or 180 days after the last chemotherapy dose), regardless of gender.

Exclusion Criteria:

1. Diagnosis of any malignancy other than gastric cancer within 5 years before the first dose (excluding cured basal cell or squamous cell skin cancers and/or carcinoma in situ treated with curative intent).
2. Imaging during screening shows tumors encasing major blood vessels or with significant necrosis/cavitation, posing a bleeding risk as determined by the investigator.
3. Currently participating in another interventional clinical study or received other investigational drugs or devices within 4 weeks before the first dose.
4. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years before the first dose. Replacement therapies (e.g., thyroid hormone, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatments.
5. Receiving systemic corticosteroid therapy (excluding nasal, inhaled, or other topical routes) or any other form of immunosuppressive therapy within 7 days before the first dose of the study.
6. Known history of allogeneic organ transplantation (excluding corneal transplants) or allogeneic hematopoietic stem cell transplantation.
7. Known allergy to any drug used in this study.
8. Not fully recovered from toxicity and/or complications of any prior interventions before starting treatment (i.e., ≤ Grade 1 or returned to baseline, excluding fatigue or alopecia).
9. Known history of human immunodeficiency virus (HIV) infection (i.e., positive HIV 1/2 antibodies).
10. Untreated active hepatitis B (defined as HBsAg positive with detectable HBV-DNA levels above the upper limit of normal at the study center).
11. Active HCV infection (HCV antibody positive with HCV-RNA levels above the lower limit of detection).
12. Received live vaccines within 30 days before the first dose (Day 1, Cycle 1). Note: Inactivated seasonal influenza vaccines administered by injection are allowed within 30 days before the first dose; however, intranasal attenuated live influenza vaccines are not permitted.
13. Pregnant or breastfeeding women.
14. Presence of any severe or uncontrolled systemic diseases, including:

    * Significant and symptomatic ECG abnormalities at rest that are difficult to control, such as complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmias, or atrial fibrillation.
    * Unstable angina, congestive heart failure, or chronic heart failure classified as NYHA ≥ Grade 2.
    * Any arterial thrombosis, embolism, or ischemia within 6 months before enrollment, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack.
    * Suboptimal blood pressure control (systolic BP > 150 mmHg, diastolic BP > 100 mmHg).
    * History of non-infectious pneumonitis requiring corticosteroid treatment within 1 year before the first dose, or current clinically active interstitial lung disease.
    * Active tuberculosis.
    * Any active or uncontrolled infection requiring systemic treatment.
    * Clinically active diverticulitis, intra-abdominal abscess, or gastrointestinal obstruction.
    * Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis.
    * Poorly controlled diabetes (fasting blood glucose > 10 mmol/L).
15. Any condition, illness, treatment, or abnormal laboratory value that could interfere with trial results, hinder the participant's full involvement in the study, or pose additional risks, as determined by the investigator. This includes any situation deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause, using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
AE | up to 24 months after enrollment or study close
  Number and percentage of participants with Adverse Events(any grade)

SECONDARY OUTCOMES:
Overall survival (OS) | up to 3 years
  The time interval between the start date of study drug and the date of death (any cause)
Duration of Response(DoR) | up to 12 months
  monitor the length of time patients experience a reduction in tumor size or stabilization of disease following the treatment
Disease control rate (DCR) | up to 12 months
  Disease control rate (DCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China